CLINICAL TRIAL: NCT07134985
Title: Pediatric Patients Who Leave the Emergency Department Without Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Pediatrician, Hillel Yaffe Medical Center
Other Study IDs: HYMC-0019-22-IL
Record Dates: First submitted 2025-08-04; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Leaving Without Being Seen or Treated
Keywords: Left Without Being Seen or Treated

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Left Without Being Seen or Treated: The patients who left without being seen or treated
  Interventions: Other: No intervention
- Discharged After Being Seen or Treated: The patients who were discharged after being seen or treated
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
Research Objectives:

To examine the clinical, operational, and demographic characteristics that influence the decision of patients to voluntarily leave the pediatric emergency department at Hillel Yaffe Medical Center before completing the evaluation or medical treatment.

DETAILED DESCRIPTION:
Patient departure from the Emergency Department (ED) before completing the medical procedure (LWBS - Left Without Being Seen or Treated) is a well-known phenomenon in emergency medicine and can be dangerous, with severe medical consequences, particularly when the patient is unaware of their condition or has not received the necessary treatment. The ED is responsible for treating urgent cases, and thus, a patient's decision to leave before completing the evaluation and/or receiving appropriate care can lead to serious consequences related to undiagnosed or improperly treated illnesses or injuries. In addition, the patient may not receive the necessary discharge instructions, which could negatively affect their health, worsen their condition, cause irreversible damage, increase the rate of repeated visits, and even pose a risk of mortality.

Numerous studies have focused on the adult population, but very few have addressed children. In pediatric EDs, the responsibility for the decision to leave the department rests with the parent or guardian, which underscores the unique importance of understanding the factors that contribute to this decision. A previous study conducted in the adult emergency department at Hillel Yaffe Medical Center found that a low triage level and long wait times were significant predictors of early departure.

Similar findings have been reported in studies conducted in the U.S. and Canada, where the impact of long wait times, ED overload, younger age, time of arrival, low urgency, and self-arrival without a referral from a physician were emphasized as contributing factors . Other studies pointed to sociodemographic variables such as nationality, gender, socioeconomic status, and previous instances of early departure as additional risk factors.

A unique study conducted among Indigenous communities in Canada highlighted factors such as feelings of discrimination, lack of trust, and poor communication with medical staff as influential in the decision of parents to leave before completing treatment [5]. Additionally, a qualitative study conducted in the U.S. using Q-methodology (a method for identifying subjective patterns of thinking by sorting statements based on agreement or relevance) found that parents left due to a lack of updates on their position in the queue, unclear information about wait times, feelings of helplessness in the face of the child's pain, or external pressures such as work or caring for other children.

Since the decision to leave in children is made by the parent and not the patient, understanding the characteristics, circumstances, and factors involved is crucial. In Israel, where the healthcare system is publicly funded and based on the National Health Insurance Law, which provides access to clinics within health funds or emergency centers, there are unique parameters that affect access to hospital care-such as referral by a physician or payment for self-referred visits. Therefore, it is likely that local, cultural, and organizational factors influence the phenomenon of early departure, and these should be examined in the pediatric context.

Due to the lack of qualitative and quantitative studies on the issue of early departure from pediatric emergency departments, both globally and particularly in Israel, there is a need to complete research aimed at filling this knowledge gap. The main reason for conducting this research is the desire to identify recurring patterns and characteristics that predict early departure, which will enable early interventions that improve service quality, reduce the risk of early departure, and decrease the medical complications resulting from it. Additionally, this study may contribute to understanding the parents' perspectives, the relationship between parents' experiences in the ED and medical decision-making, and serve as a basis for future research, training medical staff, and improving the patient and caregiver experience alike.

Research Objectives:

To examine the clinical, operational, and demographic characteristics that influence the decision of patients to voluntarily leave the pediatric emergency department at Hillel Yaffe Medical Center before completing the evaluation or medical treatment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 0-17 who arrived at the pediatric emergency department between January 2024 and December 2025.

Exclusion Criteria:

* None

Max Age: 17 Years | Sex: All
Age Groups: Child
Study Population: Children aged 0-17 who arrived at the pediatric emergency department between January 2024 and December 2025.
Sampling Method: Non-Probability Sample
Enrollment: 33000 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Descreption of the population | 1 year
  Descreption of the population of those who left without treatment in epidemiological terms.

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No
Parivate data can not be shared by institution rules.

REFERENCES:
- [Background] Gorski JK, Arnold TS, Usiak H, Showalter CD. Crowding is the strongest predictor of left without being seen risk in a pediatric emergency department. Am J Emerg Med. 2021 Oct;48:73-78. doi: 10.1016/j.ajem.2021.04.005. Epub 2021 Apr 3. PMID 33845424
- [Background] Kappy B, McKinley K, Chamberlain J, Badolato GM, Podolsky RH, Bond G, Schultz TR, Isbey S. Leaving Without Being Seen From the Pediatric Emergency Department: A New Baseline. J Emerg Med. 2023 Sep;65(3):e237-e249. doi: 10.1016/j.jemermed.2023.05.019. Epub 2023 Jun 10. PMID 37659902
- [Background] Taylor B, Young M. Pediatric ED departmental complexity: a different approach to the concept of ED crowding. CJEM. 2022 Apr;24(3):318-324. doi: 10.1007/s43678-022-00261-9. Epub 2022 Feb 11. PMID 35146700
- [Background] Kennedy M, MacBean CE, Brand C, Sundararajan V, McD Taylor D. Review article: leaving the emergency department without being seen. Emerg Med Australas. 2008 Aug;20(4):306-13. doi: 10.1111/j.1742-6723.2008.01103.x. PMID 18782204
- [Background] Bourgeois FT, Shannon MW, Stack AM. "Left without being seen": a national profile of children who leave the emergency department before evaluation. Ann Emerg Med. 2008 Dec;52(6):599-605. doi: 10.1016/j.annemergmed.2008.03.012. Epub 2008 May 1. PMID 18450328